CLINICAL TRIAL: NCT07144293
Title: Improving Physical Ability and Cellular Senescence Elimination in HIV
Acronym: IPACE-HIV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5426
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: HIV; Frailty; Prefrail; Aging Problems
Keywords: Frailty; Prefrail; Physical Function; Aging; Senescence; Senolytic therapy
MeSH Terms: conditions — Frailty | interventions — Dasatinib; Quercetin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: D+Q (Experimental)
  Interventions: Drug: Dasatinib; Drug: Quercetin
- Arm B: Placebo (Placebo Comparator)
  Interventions: Other: Placebo - Dasatinib; Other: Placebo - Quercetin

INTERVENTIONS:
Drug: Dasatinib — Dasatinib will be administered as one 100 mg capsule.
  Arms: Arm A: D+Q
Drug: Quercetin — Quercetin will be administered as five 250 mg capsules.
  Arms: Arm A: D+Q
Other: Placebo - Dasatinib — Matching Placebo for Dasatinib will be administered as one 100 mg capsule.
  Arms: Arm B: Placebo
Other: Placebo - Quercetin — Matching Placebo for Quercetin will be administered as five 250 mg capsules.
  Arms: Arm B: Placebo

SUMMARY:
This clinical trial is a Phase II study designed to test the safety and effectiveness of a combination of dasatinib and quercetin (D+Q) in improving physical function for people with HIV who are frail or prefrail. The study will involve 80 participants, all aged 50 or older, who have been living with HIV for at least 10 years determined to meet criteria for diagnosis of frail or prefrail and are currently on a stable antiretroviral therapy with viral suppression.

Participants will be randomly assigned to one of two groups: one group will receive the D+Q treatment, and the other will receive a placebo. The treatment will be given in six cycles over 12 weeks, with participants taking the medication for two days followed by 12 days without treatment. After the 12-week treatment period, participants will be monitored for another 12 weeks to assess the long-term effects.

The study aims to determine if D+Q can improve physical function and other health outcomes in this population. Randomization will be stratified by sex and age to ensure balanced groups.

ELIGIBILITY:
Inclusion Criteria:

1. Must be an older person with confirmed diagnosis of HIV-1, defined as ≥ 50 years at study entry.
2. Must have been diagnosed with HIV at least 10 years ago, as confirmed by medical records or self-report.
3. Must be on a stable effective combination antiretroviral therapy (ART) regimen, with no changes in the regimen within 12 weeks before joining the study with 2 or more consecutive HIV-RNA levels < 50 copies/mL within 48 weeks prior to study entry.
4. Must meet one or more Fried Frailty Phenotype criteria w/in 60 days prior to entry.
5. Must have eGFR > 30 using CKD-EPI per 2021 calculation equation.

Exclusion Criteria:

1. Have used quercetin or dasatinib before.
2. Need to take medications that affect CYP3A4 or interact with dasatinib (e.g., certain HIV medications).
3. Have an active cancer (except non-melanoma skin cancer).
4. Have active liver disease with a Child Pugh score greater than 6, or other significant liver problems.
5. Are on dialysis or have had a kidney transplant.
6. Have had a heart attack, angina, stroke, or mini-stroke in the last 6 months.
7. Have a known history of pulmonary arterial hypertension or other respiratory disease requiring supplemental oxygen within 60 days before joining the study.
8. Have uncontrolled diabetes with an HgbA1c level greater than 8% within 60 days before joining the study.
9. Have substance use that might interfere with study participation, as determined by the site investigator.
10. Have had a significant illness within 60 days before joining the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-11-29 (Estimated); Study Completion 2026-11-29 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Grade 2 or higher adverse events (AEs) after initiation of study treatment. | 24 weeks
Occurrence of premature treatment discontinuations. | 24 weeks
Absolute change in gait speed on 4-meter walk. | From Week 0 to Week 12

SECONDARY OUTCOMES:
Absolute change in time to complete 5 chair stands. | From Week 0 to Week 12
Absolute change in Short Performance Physical Battery (SPPB) Total Balance Test score. | From Week 0 to Week 12
  The Short Performance Physical Battery (SPPB) Total Balance Test scores range from a minimum of 0 to a maximum of 4. Higher scores indicate better balance performance.
Absolute change in the SPPB score. | From Week 0 to Week 12
  The SPPB scores range from a minimum of 0 to a maximum of 12. Higher scores indicate better physical performance.
Absolute change in 4-meter gait speed. | From Week 0 to Week 24
Absolute change in SPPB total balance test score. | From Week 0 to Week 24
  The SPPB Total Balance Test scores range from a minimum of 0 to a maximum of 4. Higher scores indicate better balance performance.
Absolute change in SPPB score. | From Week 0 to Week 24
  The SPPB scores range from a minimum of 0 to a maximum of 12. Higher scores indicate better physical performance.
Absolute change in timed chair stands. | From Week 0 to Week 24
Absolute change in plasma senescence-associated secretory phenotype (SASP) biomarkers. | From Week 0 to Weeks 12 and 24
Absolute change in serum SASP biomarkers. | From Week 0 to Weeks 12 and 24
Absolute change in cognitive function on the AIDS Clinical Trials Group (ACTG) Neuropsychology Battery "Neuropsychological Battery" section | From Week 0 to Weeks 12 and 24
  Higher scores indicate better cognitive performance.
Absolute change in symptoms of anxiety and depression using the Patient Health Questionnaire-9 (PHQ-9) assessments | From Week 0 to Weeks 12 and 24
  The PHQ-9 scores range from a minimum of 0 to a maximum of 27. Lower scores indicate better mental health, while higher scores indicate more severe depression.
Absolute change in Veterans Aging Cohort Study (VACS) Index 2.0. | From Week 0 to Weeks 12 and 24
  The VACS Index 2.0 scores range from a minimum of 0 to a maximum of 164. Higher scores indicate a higher risk of mortality and worse health outcomes.
Absolute change in participant-reported Quality of Life (QoL) on the Patient-Reported Outcomes Measurement Information System (PROMIS) QoL measure | From Week 0 to Weeks 12 and 24
  The PROMIS QoL measure have no fixed minimum score, but scores can theoretically go as low as 0 and no fixed maximum score, but scores can theoretically go as high as 100. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Alabama CRS (Site ID: 31788), Birmingham, Alabama
  - University of California, Los Angeles CARE Center CRS (Site ID: 601), Los Angeles, California
  - UCSD Antiviral Research Center CRS (Site ID: 701), San Diego, California
  - University of California, San Francisco HIV/AIDS CRS (Site ID: 801), San Francisco, California
  - Harbor University of California Los Angeles Center CRS (Site ID: 603), Torrance, California
  - University of Colorado Hospital CRS (Site ID: 6101), Aurora, Colorado
  - Whitman-Walker Institute, Inc. CRS (Site ID: 31791), Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS (Site ID: 5802), Atlanta, Georgia
  - Northwestern University CRS (Site ID: 2701), Chicago, Illinois
  - Massachusetts General Hospital CRS (MGH CRS) (Site ID: 101), Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS (Site ID: 107), Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS (Site ID: 2101), St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS (Site ID: 31786), Newark, New Jersey
  - Weill Cornell Chelsea CRS (Site ID: 7804), New York, New York
  - Columbia Physicians & Surgeons (P&S) CRS (Site ID: 30329), New York, New York
  - Weill Cornell Uptown CRS (Site ID: 7803), New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (Site ID: 31787), Rochester, New York
  - Chapel Hill CRS (Site ID: 3201), Chapel Hill, North Carolina
  - Greensboro CRS (Site ID: 3203), Greensboro, North Carolina
  - Cincinnati CRS (Site ID: 2401), Cincinnati, Ohio
  - Case CRS (Site ID: 2501), Cleveland, Ohio
  - Ohio State University CRS (Site ID: 2301), Columbus, Ohio
  - Penn Therapeutics CRS (Site ID: 6201), Philadelphia, Pennsylvania
  - University of Pittsburgh CRS (Site ID: 1001), Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics (VT) CRS (Site ID: 3652), Nashville, Tennessee
  - Houston Advancing Research Team CRS (Site ID: 31473), Houston, Texas
  - University of Washington Positive Research CRS (Site ID: 1401), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the ACTG (Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections) by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG (Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections).
  * For what types of analyses? To achieve aims in the proposal approved by the ACTG.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data.